CLINICAL TRIAL: NCT03308383
Title: Normal Echocardiographic Parameters of Indian Population and Comparison With the ASE Reference Range
Acronym: TTE IN INDIAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ganesh Kumar Munirathinam, Principal Investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NK/3908/Study
Record Dates: First submitted 2017-09-27; First posted 2017-10-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: HEALTHY

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRANSTHORACIC ECHOCARDIOGRAM (Experimental): Individuals who visit pre-anaesthetic check up (PAC) clinic for minor surgery which includes plastic, rhino-otolaryngeal, ophthalmologic, orthopaedic, abdominal, urological, gynaecological surgeries, who are free of cardiac disease or any known risk factors for the cardiac disease like chronic alcoholism, chronic smoking, metabolic syndrome, morbid obesity
  Interventions: Other: DOING TRANSTHORACIC ECHOCARDIOGRAM

INTERVENTIONS:
Other: DOING TRANSTHORACIC ECHOCARDIOGRAM — TRANSTHORACIC ECHOCARDIOGRAM WILL BE DONE IN THE PARTICIPANTS WHICH IS NON-INVASIVE

SUMMARY:
Echocardiography forms one of the most used modality in the evaluation of cardiac anatomy and functions in both patients with cardiac symptoms and in healthy individuals for occupational and research purpose. The interpretation of any medical investigation including echocardiographic report is based on its comparison with the normal range for that parameter, which is known to vary depending on the age, sex, body surface area (BSA), ethnicity and race. Since most of the medical/surgical treatment decisions are made based on the echocardiographic reports, the interpretation of results should be accurate. Even though there are many studies defining reference ranges of echocardiographic parameters, most of them were based on studies conducted in Western and European population, who shows considerable difference in their anthropometric measurements from the Indian population. Hence for the accurate diagnosis of any cardiac abnormalities, the reference values should have been derived from studies conducted in population of that particular race and ethnicity who are free of risk factors for the cardiac disease. Hence the investigator planned to conduct a study to determine the normal Echocardiographic parameters and compare it with the reference range of established by American society of echocardiography (ASE).

DETAILED DESCRIPTION:
Aim To determine the mean and standard deviation for Echocardiographic 2 dimensional, Doppler and strain parameters in Indian population and compare it with the reference range established by ASE

Materials and Methods After getting ethical clearance and informed patient consent, the study will be performed in 150 individuals who visit pre-anaesthetic check up (PAC) clinic for minor surgery which includes plastic, rhino-otolaryngeal, ophthalmologic, orthopaedic, abdominal, urological, gynaecological surgeries, who are free of cardiac disease or any known risk factors for the cardiac disease like chronic alcoholism, chronic smoking, metabolic syndrome, morbid obesity. The duration of study will be from October 2017 to June 2018 or till 150 individual studied.

Echocardiographic Study For all the individual electrocardiogram (ECG) integrated TTE will be done using general electric (GE) Echocardiographic machine using the cardiac probe of frequency 5 Hz in supine or left lateral position in a comfortable environment. All images will be recorded as per the ASE recommendations and the images will be analysed by echo cardiographer accredited by the national board of echocardiography. Three consecutive cardiac cycles were measured and average of the three will be taken for analysis.

Image acquisition By placing the Transducer in the left third or fourth intercostal space adjacent to the sternum parasternal short axis (PSAX) view is obtained, by tilting the probe superiorly and inferiorly, the true short axis view of the LV where both the papillary muscle are seen. Parasternal long axis (PLAX) view is formed by rotating the probe perpendicular from the true PSAX view. By applying M mode across the tip of the MV in PLAX view the end diastolic, end systolic dimensions of LV, posterior wall and inter-ventricular septum thickness, relative wall thickness (RWT) and LV internal dimension will be measured from leading edge to leading edge.1 From the same image FS, LVEF by Teicholtz method, LV mass by linear cube method will be calculated.

LV EF (Teicholtz)32 :

LVEDV = 7/(2.4+LVEDD) X LVEDD3 LVESV = 7/(2.4+LVESD) X LVESD3 LV FS32 = (LVEDD-LVESD/LVEDD) x 100 LV mass in grams = 0.8x{1.04x[(IVSd+PWd+LVEDD)3 - LVIDD3]} +0.6.1 RWT = (2 X PW thickness)/ LVEDD.33

By moving the transducer cranially and medially towards sternum, and by placing M mode across the aortic sinus, perpendicular to the long axis of the aorta, LA AP diameter will be measured from leading edge to leading edge at the end of systole. From the same 2D image the aortic annulus, sino-tubular junction (STJ), aortic sinus and ascending aorta diameter will be measured from leading edge to leading edge.1 By tilting the probe from the PLAX view towards the sternum, the distal RVOT will be in view and diameter of which is measured from the leading edge to the leading edge. Proximal RVOT diameter is measured from the leading edge to the leading edge at the diastole in PSAX view in which the right ventricular (RV) inflow and outflow is visible,31 in the same view the diameter of the pulmonary valve (PV) annulus will be measured.

On palpation, the apical impulse will be identified and by placing the transducer in that point with the probe pointing toward the right shoulder, apical 4 chamber (A4C) view is obtained. The image will be optimized to get the maximum length of the LV to avoid foreshortening by identifying the pinching apex. LV end systolic volume (LVESV) and EDV and EF will be measured by Simpson's method. And by applying pulse wave Doppler with the sample volume at the tip of the mitral leaflet, mitral valve E, A velocity and deceleration time and A wave duration are calculated.

In the same image by applying Tissue Doppler (TDI) over mitral valve lateral and septal annulus e', a', S', TEI index, isovolumic relaxation time (IVRT) and isovolumic contraction time (IVCT) are calculated. TEI index is calculated using the formula (IVRT+IVCT)/ET, where ET is the ejection time. By applying M mode across the lateral annulus of the MV, mitral annular plane systolic excursion (MAPSE) is measured in cms. All the Doppler measurement will be done with the acceptable alignment between the cursor angle and movement of the tissue or blood flow (<20 degree).

Strain will be measured for both the lateral and septal wall of the LV in the same image.

By tilting the probe towards sternum and bringing the TV in the focus, the apical RV focussed view is formed. TV annulus, RV basal and mid diameter and the RV length are measured from the leading edge to the leading edge. And by applying TDI at the lateral annulus of TV e', a', s', TEI index are measured. On applying M mode across the lateral annulus, tricuspid annular plane systolic excursion (TAPSE) is measured. FAC which is measured by {RV diastolic area (DA) - RV systolic area (SA)}/ RV DA, and RV lateral wall strain are measured.

Subcostal view is obtained by placing the probe in the xiphi-sternum directing towards the left shoulder. Patient can be asked to flex the legs to make the abdominal wall relax for the placement of the probe. The RV lateral wall thickness and TV annulus diameter is measured in the subcostal 4 chamber view. And on placing the probe vertically with the pointer directed cephalad the inferior vena cava (IVC) is seen in the long axis which can be used for measuring the IVC diameter at the end expiration.

All measurements were divided by BSA for the indexed measurements. The peak of R wave and the beginning of the T wave in the ECG are used to identify the end of diastole and end of systole respectively while performing measurement.

ELIGIBILITY:
Inclusion Criteria:

- Age between18 to 60 years

Exclusion Criteria:

* History of congenital or acquired cardiac abnormality
* Symptoms and Signs suggestive of any cardio-respiratory disease
* Systemic hypertension SBP more than 140 and DBP more than90
* Known case of Diabetes mellitus or signs and symptoms suggesting like polyuria, polydipsia, autonomic dysfunction
* History of long term exercise
* Systemic disease like chronic kidney disease, chronic liver disease, chronic obstructive pulmonary disease
* LVH or any abnormality in ECG
* Abnormal chest X-ray
* Obesity defined by BMI MORE THAN 25 kg/m2)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
EDLVID | up to 30 minutes
  End diastole left ventricle internal diameter
ESLVID | up to 30 minutes
  End systole left ventricle internal diameter
EDIVST | up to 30 minutes
  End diastole inter-ventricular septum thickness
ESIVST | up to 30 minutes
  End systole inter-ventricular septum thickness
EDPWT | up to 30 minutes
  End diastole posterior wall thickness
ESPWT | up to 30 minutes
  End systole posterior wall thickness
LVEF | up to 30 minutes
  Left ventricle ejection fraction
LV strain | up to 30 minutes
  Left ventricle strain
TAPSE | up to 30 minutes
  Tricuspid annular plane systolic excursion
RV FAC | up to 30 minutes
  Right ventricle fractional area change
RV TEI index | up to 30 minutes
  Right ventricle TEI index
Mitral and tricuspid E',A', S' | up to 30 minutes
  Mitral and tricuspid annular tissue velocities
RVOT diameter | up to 30 minutes
  Right ventricle outflow tract diameter
Mitral tricuspid aortic pulmonary annulus diameter | up to 30 minutes
  Mitral tricuspid aortic pulmonary annulus diameter

CONTACTS AND LOCATIONS:
Overall Officials: GANESH KUMAR, MD, Principal Investigator — PGIMER, CHANDIGARH, INDIA
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No